CLINICAL TRIAL: NCT01922596
Title: Effect of Adductor Canal Blockade vs Femoral Nerve Blockade on Muscle Strength, Mobility and Pain in Patients With Severe Pain After Total Knee Arthroplasty
Brief Title: Adductor Canal Blockade vs Femoral Nerve Blockade on Muscle Strength, Mobility and Pain After TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Ulrik Grevstad, Consultant, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM3_UG_12; 2012-004554-28 (EudraCT Number)
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Mobility After Total Knee Arthroplasty
Keywords: Total Knee Arthroplasty; Adductor Canal Blockade; Us-guided nerve blockade
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active FNB, placebo ACB (Experimental): FNB with 30 ml of ropivacaine 0,2% and ACB with 30 ml of placebo (saline). The ACB will be performed just prior to the FNB. The blockades will be performed just after obtaining the baseline values (outcome measures) at time 0.
  Interventions: Drug: Ropivacaine; Drug: Placebo
- Active ACB, placebo FNB (Experimental): ACB with 30 ml of ropivacaine 0,2% and FNB with 30 ml of placebo (saline.The ACB will be performed just prior to the FNB. The blockades will be performed just after obtaining the baseline values (outcome measures) at time 0.
  Interventions: Drug: Ropivacaine; Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine
  Other Names: Naropin
Drug: Placebo
  Other Names: Saline

SUMMARY:
The purpose of the study is to compare the effect of a Adductor Canal Blockade (ACB) vs a Femoral Nerve Blockade (FNB), on muscle strength, mobility and pain in patients with severe pain (VAS pain score > 60) after Total Knee Arthroplasty (TKA.

DETAILED DESCRIPTION:
The patients will be included after surgery (the first 2 postoperative days). Patients reporting VAS > 60 during active flexion of the knee can be included. All included patients will receive 2 blockades at the same time - an ACB and a FNB, one blockade with 30ml ropivacaine 0,2% and the other with 30ml saline according to randomization.

Prior to, and after, the blockades VAS pain scores will be obtained, muscle strength (quadriceps and adductors) will be measured using a handheld dynanometer and a Timed Up and Go test will be performed.

The study is registered at clinicaltrials.gov after inclusion of the first patient. The reason for this is that we recently became aware of that some journals do not accept a EudraCT registration. The study was registered at EudraCT (2012-004554-28)prior to enrollment of patients.

ELIGIBILITY:
Inclusion Criteria:

* TKA within 72 hours and VAS>60 during 45 degrees active flexion of the knee despite conventional pain medication
* informed consent
* ASA 1-3
* BMI 18-40

Exclusion Criteria:

* Unable to communicate in Danish
* Allergic reactions toward ropivacaine
* Alcohol and or drug abuse
* Unable to cooperate
* Known sensory disturbances in the lower limbs

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change i muscle strength of the quadriceps muscle, after the blockade | 0 and 120 minutes
  Maximum Voluntary Isometric Contraction (MVIC) of the quadriceps femoris muscle will be measured before and 2 hours after the blockade. The change will be compared between the groups. At each measuring point three measurements will be made and the average of these used.

SECONDARY OUTCOMES:
muscle strength, adductor muscles | 0 and 120 minutes
  MVIC of the adductors will be measured before and 2 hours after the blockades. The change will be compared between the groups. At each measuring point three measurements will be made and the average of these used.
Timed Up and Go (TUG)test | 0 and 120 minutes
  The change in time to perform a TUG test before and after the blockades will be compared between the groups. Also the change in highest pain score during the TUG tests will be compared between the groups
VAS pain scores at rest | 0 and 120 minutes
  VAS pain scores at rest will be obtained before VAS pain scores during passive flexion of the knee.
  The change between groups will be compared
Pain during passive flexion of the knee | 0 and 120 minutes
  VAS pain scores during passive 45 degrees flexion of the knee. The change will be compared between the groups. VAS during passive flexion will be obtained prior to the MVIC measurements and the TUG test

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Grevstad, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Grevstad U, Mathiesen O, Valentiner LS, Jaeger P, Hilsted KL, Dahl JB. Effect of adductor canal block versus femoral nerve block on quadriceps strength, mobilization, and pain after total knee arthroplasty: a randomized, blinded study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):3-10. doi: 10.1097/AAP.0000000000000169. PMID 25376972